CLINICAL TRIAL: NCT01768988
Title: Efficacy Of Pregabalin In The Treatment Of Pancreatic Cancer Pain. A Randomized Controlled Double-Blind, Parallel Group Study
Acronym: PANPAIN/1
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Change of PI. Former PI changed from Research Center and Promoter obliged unexpectedly to change the PI.
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, CDursteler, MD, PhD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PANPAIN/1
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Pancreatic Cancer; Visceral Pain
MeSH Terms: conditions — Pancreatic Neoplasms; Visceral Pain | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I (Experimental): Conventional analgesic treatment + pregabalin.
  Interventions: Drug: Pregabalin
- Group II (Placebo Comparator): Conventional analgesic treatment + placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Conventional treatment + placebo (during 90 days).
  Conventional treatment comprises a WHO step ladder approach and comprises in most cases:
  1. Paracetamol 1g/8h
  2. Weak opioid (tramadol at maximal doses of 400 mg/24h)
  3. Strong opioid in substitution of weak opioid if not efficient (e. g. morphine, oxycodone, fentanyl patch, hidromorphone), at the needed doses to control pain (VAS < 3).
  Arms: Group II
Drug: Pregabalin — Treatment during 90 days with conventional treatment + pregabalin.
  Pregabalin doses were reached until the maximal doses (300 mg/12h) depending on patient tolerability. An escalating dose scheme were desigened as follows, to avoid tolerability problems:
  Week 1 75-0-75 Week 2 75-0-150 Week 3 150-0-150 Week 4 150-0-300 Week 5 300-0-300 (until the end of study)
  Conventional treatment comprises a WHO step ladder approach and comprises in most cases:
  1. Paracetamol 1g/8h
  2. Weak opioid (tramadol at maximal doses of 400 mg/24h)
  3. Strong opioid in substitution of weak opioid if not efficient (e. g. morphine, oxycodone, fentanyl patch, hidromorphone), at the needed doses to control pain (VAS < 3).
  Arms: Group I

SUMMARY:
This is a randomized, double blind controlled, parallel arms trial, aimed to assess the efficacy of pregabalin on pancreatic cancer induced abdominal pain. The goals of this study include (1) assessing the analgesic effect of pregabalin in comparison to placebo; assessing the presence of central sensitization and its potential reversion by Pregabalin; (3) assessing quality of life of patients treated with pregabalin in comparison to placebo; (4) to compare adverse effects in patients treated with Pregabalin in comparison to placebo; (5) to compare anxiety and depression in patients treated with pregabalin in comparison to placebo.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients > 18 years old recently diagnosed of pancreatic cancer (<3 months).
* 2. Personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the trial.
* 3. Patients willing and able to comply with the scheduled visits, treatment plan, laboratory tests and other trial procedures.

Exclusion Criteria:

* 1. Patients with evidence or history of medical or surgical disease of importance for this study as judged by investigator.
* 2. Patients with previously diagnosed moderate to severe renal impairment. Those with a Clearance of Creatinine (CLcr) < 60mL/min should be excluded.
* 3. Patients treated with anticonvulsants during the previous 4 months.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-08; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity (Visual Analogue Scale; VAS Score) | From baseline to day 90.
  Analgesic effect of pregabalin therapy in pancreatic cancer patients, assessed using a visual analogue scale (VAS), the Brief Pain Inventory (BPI) and Neuropathic Pain VAS score.

SECONDARY OUTCOMES:
Quality of life | From baseline to day 90.
  Changes in quality of life compared to baseline level using SF-36 (Short-Form Health Survey) quality of life questionnaire.
Performance status | From baseline until to day 90.
  Performance status (Karnofsky Performance Status Scale).
Anxiety and depression | From baseline to day 90.
  Anxiety and depression will be also assessed, using Hospital Anxiety and Depression Scale (HADS).
Neuropathic Pain | From baseline to day 90.
  Neuropathic pain participation will be measured by a neuropathic pain questionnaire (NPSI).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Spain